CLINICAL TRIAL: NCT06306508
Title: Investigation of the Effect of Parental Illness Beliefs and Anxiety Level on Functional and Physical Level of the Child in Children With Cystic Fibrosis
Brief Title: Effect of Parental Attitude on Functional and Physical Level of Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Asst. Prof., Halic University
Other Study IDs: HUvbayraktaroglu
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis in Children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some parents may be more protective of children with CF due to concerns about worsening of the disease due to infection, which can affect their functional level. The goal of this observational study is to learn about the family's protective approach to the functioning and disease course of children with cystic fibrosis (CF) to determine whether there are possible negative effects. There will be an alternative viewpoint offered to clinicians regarding the management of CF with outputs of this study.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an inherited disease characterized by pulmonary involvement. Children with CF may have low levels of physical activity, physical fitness and functional capacity, and peripheral muscle weakness. Parents who take care of children with CF may be protective of their children's social environment due to reasons such as the risk of infection. Based on the idea that parents may have potential limitations on their children with CF, the aim of this study was to examine the effect of parental illness beliefs and anxiety levels on the functional and physical level of the child. Children with CF will be administered Modified Shuttle Walking Test, Munich Physical Fitness Test, quadriceps muscle strength and hand grip strength test, respiratory function and respiratory muscle strength test, Child Physical Activity Questionnaire, Shortness of Breath Beliefs Questionnaire, Revised Cystic Fibrosis Questionnaire, Parental Attitude Scale, Perceived Social Support Scale. Parents will be administered the Shortness of Breath Beliefs Questionnaire (Parent version), Revised Cystic Fibrosis Questionnaire (Parent version), Parent Attitude Scale, Fear of Disease Progression Questionnaire for Parents. The level of correlation between the outcomes of the scales administered to parents and the assessment outcomes administered to children will be examined.

ELIGIBILITY:
* Inclusion Criteria:

  1. For a child

     1. To be between 7-17 years old,
     2. Living with family or caregiver.
  2. For the parent

     1. Being the mother, father or other caregiver of the child,
     2. Voluntarily agreeing to participate in the study on behalf of both the child and oneself.
* Exclusion Criteria:

  1. For the child

     1. Having cognitive impairment that would prevent participation in the study or being able to cooperate with the measurements and not being able to adapt,
     2. History of previous lung or liver transplantation,
     3. History of hospitalization within the last 1 month,
     4. Having a neurological or orthopedic comorbidity that affects mobility.
  2. For the parent

     1. Having cognitive impairment at a level that prevents participation in the study
     2. Not living in the same household with the child.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cystic fibrosis and their parents who visited a private hospital's Pediatric Chest Diseases Outpatient Clinic made up the study's population. 37 parents of children with cystic fibrosis and their 37 offspring who match the inclusion and exclusion criteria and willingly consent to take part in the study will make up the sample.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Modified shuttle walk test (MST) | only baseline
  Functional capacity

SECONDARY OUTCOMES:
Forced expiratory volume at one second (FEV1) | only baseline
  It is being evaluated to assess lung function. A spirometry is used for the assessment.
Forced vital capacity (FVC) | only baseline
  It is being evaluated to assess lung function. A spirometry is used for the assessment.
Forced expiratory volume at one second / Forced vital capacity rate (FEV1/FVC) | only baseline
  It is being evaluated to assess lung function. A spirometry is used for the assessment.
Peak expiratory flow (PEF) | only baseline
  It is being evaluated to assess lung function. A spirometry is used for the assessment.
Maximum inspiratory pressure (MIP) | only baseline
  It is being evaluated to assess inspiratory muscle strength. A intraoral pressure meter device is used for the assessment.
Maximum expiratory pressure (MEP) | only baseline
  It is being evaluated to assess expiratory muscle strength. A intraoral pressure meter device is used for the assessment.
Physical Activity Questionnaire for Children (PAQ-C) | only baseline
  The PAQ-C is a scale that assesses moderate to vigorous physical activity over the past seven days. For each item of the questionnaire, except for the tenth question that inquires about the disease status, an evaluation is made on a 5-point scale and an activity score between 1-5 is found. After the scores of the answers given to the nine questions are summed and divided by the number of questions, the score obtained is the total physical activity score of the child from the questionnaire. An average score of "1" indicates a low level of physical activity, while an average score of "5" indicates high physical activity.
Munich physical fitness test (MFT) | only baseline
  The test consists of six parameters: ball bounce, target catch, forward bending, vertical jump, hang and step test. With this test, peer comparison according to age and gender and interpretation of motor performance can be made with objective scores. The total fitness score is the average of the six parameter scores. Physical fitness is classified as inadequate (≤35), normal (36-45), adequate (46-55), good (56-65) or very good (≥66) according to the total score.
Quadriceps strength | only baseline
  It is being evaluated to assess quadriceps muscle strength. A hand-held dynamometer is used for the assessment.
Handgrip strength | only baseline
  It is being evaluated to assess handgrip strength. A hand dynamometer is used for the assessment.
Cystic Fibrosis Questionnaire Revised (CFQ-R) | only baseline
  The CFQ-R assesses quality of life. The CFQ-R is a cystic fibrosis-specific scale developed separately for both the child and the parent. Both versions are used in this study. The child version of the questionnaire consists of 35 items and the parent version consists of 50 items. Scores for each HRQoL domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health. CD-Rom Program available for scoring the CFQ-R.
Parental Attitude Scale (PAS) | only baseline
  The PAS was developed to measure parents' child-rearing attitudes. Democratic (17 items), Authoritarian (11 items), Overprotective (9 items), Permissive (9 items). In scoring, scores and corresponding responses were 5 for "always", 4 for "most of the time", 3 for "sometimes", 2 for "rarely" and 1 for "never". Having a high score meant to adopt the behavior style represented by that domain.
Parent Attitude Scale | only baseline
  The scale has three sub-dimensions: acceptance/affection, control/supervision and psychological autonomy. Accordingly, since the scale is scored as Always 5; Mostly 4; No opinion 3; Occasionally 2; Never 1, the individual to whom the scale is applied receives a minimum score of 15 and a maximum score of 75 from each dimension separately. Each dimension is evaluated according to whether the scores are low or high. In whichever dimension the score is higher, it is accepted that the child perceives parental attitude in that way.
Perceived Social Support Scale (PSS) | only baseline
  PSS was developed to measure the social support perceived by children. The scale includes 5 items on social support perceived from mother and 5 items on social support perceived from father, and 4 items on social support perceived from peers. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. As the total score increases, the child's perception of social support increases.
Breathlessness Beliefs Questionnaire (BBQ) | only baseline
  The questionnaire was developed based on the Tampa Kinesiophobia Scale to assess patients' dysfunctional beliefs about dyspnea due to reduced physical activity. The items question the patient's beliefs about the effects of dyspnea and whether activity should be avoided. The questionnaire has a minimum score of 11 and a maximum score of 55. As the total score increases, the belief in dysfunctional dyspnea increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Haliç University, Istanbul, Eyup, Turkey (Türkiye)